CLINICAL TRIAL: NCT00005463
Title: Population-Based Modeling of Cholesterol Lowering in the United States
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4907; R01HL046315 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2002-09

CONDITIONS: Cardiovascular Diseases; Coronary Heart Disease Risk Reduction; Heart Diseases; Coronary Disease; Hypercholesterolemia
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Hypercholesterolemia

SUMMARY:
To evaluate the cost-effectiveness of cholesterol-lowering strategies in the United States population. The study used the Coronary Heart Disease (CHD) Policy Model, a state-transition computer simulation model used to obtain forecasts of the public health impact and economic cost of CHD in the United States population.

DETAILED DESCRIPTION:
BACKGROUND:

The study was part of an Institute-initiated Request for Applications (RFA) titled "Cost-Effective Strategies of Cholesterol-Lowering" released by the NHLBI in 1990. The RFA was stimulated by the controversy concerning costs and cost-effectiveness that followed the 1987 report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults. The RFA was intended to support a broad and thorough quantitative exploration of the potential health benefits and costs of cholesterol-lowering from multiple perspectives.

DESIGN NARRATIVE:

The study added to the CHD Policy Model the capability to model the consequences of reductions in LDL cholesterol and increases in HDL/LDL ratios in the United States population. The CHD Policy Model was used for several studies, including: to compare the implications of using alternative epidemiologic studies as the basis for estimating the association between cholesterol levels and CHD risk; to derive cutting points for initiating cholesterol reduction, specific to age, sex, and CHD risk factors, and based on cost-effectiveness criteria; to compare the cost-effectiveness of specific targeted and population-wide strategies for cholesterol reduction; to incorporate the effects of treatments on quality of life, including both adverse effects of cholesterol-lowering drugs and reductions in CHD morbid events; and finally, to perform a cost-effectiveness analysis of cholesterol screening, incorporating costs of screening, effects of measurement error on misclassification of patients, and variations in individual cholesterol levels over time.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-08; Study Completion 1993-05 (Actual)

REFERENCES:
- [Background] Goldman L, Goldman PA, Williams LW, Weinstein MC. Cost-effectiveness considerations in the treatment of heterozygous familial hypercholesterolemia with medications. Am J Cardiol. 1993 Sep 30;72(10):75D-79D. doi: 10.1016/0002-9149(93)90015-5. PMID 8213502
- [Background] Hunink MG, Goldman L, Tosteson AN, Mittleman MA, Goldman PA, Williams LW, Tsevat J, Weinstein MC. The recent decline in mortality from coronary heart disease, 1980-1990. The effect of secular trends in risk factors and treatment. JAMA. 1997 Feb 19;277(7):535-42. PMID 9032159
- [Background] Tosteson AN, Weinstein MC, Hunink MG, Mittleman MA, Williams LW, Goldman PA, Goldman L. Cost-effectiveness of populationwide educational approaches to reduce serum cholesterol levels. Circulation. 1997 Jan 7;95(1):24-30. doi: 10.1161/01.cir.95.1.24. PMID 8994412